CLINICAL TRIAL: NCT02047175
Title: A Randomized, Open-label, Multiple-dose, Two-arm, One-sequence • Crossover Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration Telmisartan/S-amlodipine and Rosuvastatin in Healthy Volunteers
Brief Title: CKD-346 DDI Study(Telmisartan/S-Amlodipine, Rosuvastatin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 147DDI13019
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(Telmisartan/S-Amlodipine) (Experimental): A(Telmisartan/S-Amlodipine)
  : Telmisartan/S-Amlodipine 40/2.5mg 2T for 9days and Telmisartan/S-Amlodipine 40/2.5mg 2T + Rosuvastatin 20mg 1T for 5days
  Interventions: Drug: Telmisartan/S-Amlodipine; Drug: Telmisartan/S-Amlodipine + Rosuvastatin
- B(Rosuvastatin) (Experimental): B(Rosuvastatin)
  : Rosuvastatin 20mg 1T for 5days and Telmisartan/S-Amlodipine 40/2.5mg 2T + Rosuvastatin 20mg 1T for 9days
  Interventions: Drug: Rosuvastatin; Drug: Telmisartan/S-Amlodipine + Rosuvastatin

INTERVENTIONS:
Drug: Telmisartan/S-Amlodipine — Telmisartan/S-Amlodipine 40/2.5mg 2T PO, QD for 9days
  Other Names: Telminuvo tablet
  Arms: A(Telmisartan/S-Amlodipine)
Drug: Rosuvastatin — Rosuvastatin 20mg 1T PO, QD for 5days
  Other Names: Crestor tablet
  Arms: B(Rosuvastatin)
Drug: Telmisartan/S-Amlodipine + Rosuvastatin — Telmisartan/S-Amlodipine 40/2.5mg 2T + Rosuvastatin 20mg 1T PO, QD for 5days
  Other Names: Telminuvo tablet + Crestor tablet
  Arms: A(Telmisartan/S-Amlodipine)
Drug: Telmisartan/S-Amlodipine + Rosuvastatin — Telmisartan/S-Amlodipine 40/2.5mg 2T + Rosuvastatin 20mg 1T PO, QD for 9days
  Other Names: Telminuvo tablet + Crestor tablet
  Arms: B(Rosuvastatin)

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction of CKD-346(Telmisartan/S-Amlodipine, Rosuvastatin)

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, two-arm, one-sequence · crossover study to evaluate the safety and pharmacokinetics after oral concurrent administration telmisartan/s-amlodipine and rosuvastatin in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female between 20 and 45 years of age (inclusive) at the pre-study (screening)
2. Participant who has a body weight that is >55kg(male) or >50kg(female) with ideal body weight of 80-120% (ideal body weight) = {Height(cm) - 100} * 0.9
3. If female, must include more than one among the items

   1. The menopause (there is no natural menses for at least 2 years)
   2. Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition)
   3. The male partner infertility before screening (Demonstrated azoospermia after vasectomy)and if this man is the only partner of the female subject.
   4. you are using one of the following contraceptive measure for 3 months before screening, and Necessarily you agree that used continuously contraceptive measure during the clinical trial and for 1 month after the final dosing investigational product.(But, should not use a device of contraception or oral contraceptive drug that containing a hormonal caused telmisartan, s-amlodipine, atorvastatin calcium drug interactions during the clinical trials)

      * Abstinence.
      * Physical interrupt method (such as a condom, contraceptive diaphoretic or cervical cap)
   5. In case of women of childbearing age, the serum β-hCG pregnancy test is negative before taking the investigational product, and urine β-hCG test is negative before taking the investigational product.
4. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms during clinical trials and do not sperm donation during clinical trials and until one month after the final dosage of investigational products
5. Those who fully understand about this clinical trial after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent.

Exclusion Criteria:

1. The subject has a previous history of any clinically significant cardiovascular, pulmonary, renal, endocrine, hematological, gastro-intestinal, neurological, psychiatric, or malignancy.
2. Have a gastrointestinal disease history that can affect drug absorption (Crohn's disease, ulcers, etc.) or surgery (except simple appendectomy or hernia surgery).
3. Hypersensitivity reaction to drug or clinically significant hypersensitivity reaction in the history of Investigational drugs (telmisartan, s-amlodipine or rosuvastatin calcium) or additives.
4. An impossible one who participates in clinical trial including screening tests(medical history taking, V/S, physical examination, 12-lead ECG, blood & urine laboratory test result)
5. Defined by the following laboratory parameters:

   * Hemoglobin < 13.0 g/dL(male), Hemoglobin < 12.0 g/dL(female)
   * AST, ALT> 1.25* upper limit of normal range
   * Total bilirubin > 1.5* upper limit of normal range
   * CPK > 1.5* upper limit of normal range
   * eGFR(using by MDRD method) < 60 mL/min/1.73m2
6. Sitting SBP > 150 mmHg or < 90 mmHg, Sitting DBP> 100 mmHg or < 50 mmHg , after 5minuts break.
7. Drug abuse or have a history of drug abuse showed a positive for urine drug test.
8. Female Participant is pregnant or lactating
9. A heavy caffeine consumer(caffeine>5cups/day), alcohol consumer(alcohol>210g/week), or smoker(cigarette>10cigarettes/day)
10. Participation in any other study and have received any other investigational drug or device within 90 days prior to study treatment.
11. Administration of drug metabolizing enzyme inducers or inhibitors such as barbitals within 30 days prior to the first dosing.
12. Blood donation (1 unit or more) within 60 days prior to study treatment or plasma donation within 30 days prior to study treatment.
13. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1L per a day or more within 7 days before the beginning of study treatment)
14. Subject takes ethical drug or herbal medicine within 14days, OTC or vitamins within 7days before the beginning of study treatment.
15. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.

    -

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
AUCt,ss of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
Cmax,ss of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
AUCt,ss of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h
Cmax,ss of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h

SECONDARY OUTCOMES:
Tmax,ss of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
T1/2 of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
CL/F of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
Vd/F of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
R of Telmisartan/S-Amlodipine | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24h
Tmax,ss of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h
T1/2 of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h
CL/F of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h
Vd/F of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h
R of Rosuvastatin | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24h

CONTACTS AND LOCATIONS:
Overall Officials: Dong-seok Yim, professor, Principal Investigator — The Catholic University of Korea
Locations (1):
- The catholic university of Korea, seoul ST.Mary's hospital, Seoul, Gangnam-gu, South Korea